CLINICAL TRIAL: NCT06015945
Title: Role of Home-based Transcutaneous Electrical Acustimulation for Treatment of Pain in Patients With Chronic Pancreatitis- A Pilot Study
Brief Title: Role of Home-based Transcutaneous Electrical Acustimulation for Treatment of Pain in Patients With Chronic Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jorge Machicado, MD, MPH, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00225786
Record Dates: First submitted 2023-08-22; First posted 2023-08-29 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pancreatitis
Keywords: Abdominal pain; Transcutaneous Acustimulation
MeSH Terms: conditions — Pancreatitis, Chronic; Abdominal Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Transcutaneous Electrical Acustimulation (TEA) (Experimental)
  Interventions: Device: Transcutaneous Electrical Acustimulation (TEA)

INTERVENTIONS:
Device: Transcutaneous Electrical Acustimulation (TEA) — The severity and frequency participants pain will be measured during a run-in period of 2 weeks to assess baseline pain severity and frequency. Eligible participants will have a 4-week treatment period at home. Stimulation with the TEA device will be performed for 30 minutes twice per day, in the morning and in the evening.
  In addition to using the device, participants will have study visits, complete surveys, as well as provide medical information during the study.

SUMMARY:
This research is studying a new noninvasive device-based therapy called Transcutaneous Electrical Acustimulation (TEA) to learn about its safety and how well it works as a treatment of pain in chronic pancreatitis. The purpose of this study is to investigate the potential of TEA to treat abdominal pain in patients with chronic pancreatitis (CP).

The study hypothesizes that TEA can be used as a non-pharmaceutical opioid-free approach to treat pain in chronic pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic pancreatitis (CP), based on a score greater or equal to 4 using a previously validated Mayo scoring system that uses morphologic and functional criteria, or endosonographic features suggestive or consistent with CP based on Rosemont criteria.
* Abdominal pain present at least once within the last month
* Willing and able to provide written informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding mother
* Imprisoned individuals
* Non-English speaking patients
* Scheduled for or with a history of pancreatic surgery (e.g. Total Pancreatectomy with Islet Auto Transplantation (TPIAT), Puestow, Frey, Whipple, other)
* Currently undergoing or about to start endoscopic therapy with Endoscopic retrograde cholangiopancreatography (ERCP) or Endoscopic ultrasound (EUS)
* Recent history of acute pancreatitis as defined by the Revised Atlanta Classification within a month prior to enrollment
* Radiologic and clinical findings consistent with symptomatic pseudocyst, wall-off necrosis, infected pancreatic necrosis, or biliary obstruction within the last 6 months
* Self-reported daily use of opioids for > 12 months for weak opioids (codeine, tramadol and hydrocodone) or > 6 months for strong opioids (other opioids) in the last two years.

-Self-reported ongoing illicit drug use or abuse-

* Suspected or diagnosed pancreatic cancer
* Receiving chemotherapy for cancer
* Known allergy to adhesive electrocardiogram (ECG) electrodes
* Patients with bilateral below the knee amputation
* Patients with lower extremity paralysis
* Patient is participating in another clinical trial
* Patients with an implantable electrical stimulation device.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Machicado, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two consented, potentially eligible individuals did not complete the run-in period and, therefore, were determined to not be eligible to become participants.
Period: Overall Study
Arm/Group | Transcutaneous Electrical Acustimulation (TEA)
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Baseline data was collected from all participants who were consented and, at the end of the 2-week run-in period, remained eligible to begin the trial.
Arm/Group | Transcutaneous Electrical Acustimulation (TEA)
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Approached Individuals Who Met Eligibility Criteria
Description: This feasibility outcome measured eligibility of individuals to participate, as opposed to any effects of the intervention. Results reflect the total number of individuals who were approached as the number analyzed, and of that population, the number who were eligible to be consented and proceed to the run-in period.
Time Frame: Approximately 1 year (during the recruitment period)
Population: NOTE: 178 individuals were approached to determine whether they were eligible to participate in this trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Transcutaneous Electrical Acustimulation (TEA)
Number analyzed (Participants) | 178
Participants | 12

2. Primary Outcome: Proportion of Approached and Eligible Participants Who Provided Informed Consent
Description: This outcome measured feasibility and willingness of individuals to participate, as opposed to any effects of the intervention. Therefore, the "participants" analyzed below include all of the individuals determined to be eligible as shown in Outcome Measure 1.
Time Frame: Approximately 1 year (during the recruitment period)
Population: All "participants" included in this outcome measure provided informed consent regardless of whether they completed the run-in period, which would allow them to proceed to become participants in the actual trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Transcutaneous Electrical Acustimulation (TEA)
Number analyzed (Participants) | 12
Participants | 12

3. Primary Outcome: Proportion of Participants Who Met the Eligibility Criteria After the run-in Period for the Participants Who Provided Informed Consent.
Description: This outcome measured feasibility and continued eligibility of individuals to allow them to begin to participate in the actual trial, as opposed to any effects of the intervention. Therefore, the "participants" analyzed below include all of the individuals who were determined to be eligible and who were consented, as shown in Outcome Measure 2. These "participants" began a 2-week run-in period to confirm baseline pain and trial eligibility. Results reflect participants who were determined to still be eligible after the run-in period.
Time Frame: Approximately 2 weeks
Population: "Participants" analyzed in this outcome measure provided informed consent, even though some of them were subsequently determined to be ineligible at the end of the run-in period to participate in the actual trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Transcutaneous Electrical Acustimulation (TEA)
Number analyzed (Participants) | 12
Participants | 10

4. Primary Outcome: Proportion of Participants Who Started the Intervention Among Those Who Met run-in Period Criteria.
Description: Results reflect the participants who completed the run-in period and received the first TEA treatment.
Time Frame: Baseline visit (V1)
Measure: Count of Participants; unit: Participants
Arm/Group | Transcutaneous Electrical Acustimulation (TEA)
Number analyzed (Participants) | 10
Participants | 9

5. Primary Outcome: Proportion of Participants That Adhere to the Intervention as Prescribed Among Participants That Start the Intervention
Description: Adherence will be directly monitored through use of the TEA device. The TEA automatically records duration of use, time of the day, and stimulation intensity.
Time Frame: Weeks 1-4 (after the 4-week treatment period)
Population: Adherence to the duration of TEA use, times of daily use, and stimulation intensity, were supposed to be automatically recorded by the device. However, these data did not download properly in any of the devices and, as a result, all the data was unusable, so no data was collected. There are no plans to collect this data in the future.
Arm/Group | Transcutaneous Electrical Acustimulation (TEA)
Number analyzed (Participants) | 0

6. Primary Outcome: Proportion of Participants Who Completed Follow up Visit at 4 Weeks and Return Complete Follow-up Questionnaires at Week 8, Among Participants Who Started the Intervention
Description: Results reflect participants who started the TEA and who returned the follow-up questionnaires at week 4 and week 8 (end of the study).
Time Frame: Week 8
Population: 1 participant withdrew prior to starting treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Transcutaneous Electrical Acustimulation (TEA)
Number analyzed (Participants) | 9
Participants | 7

7. Primary Outcome: Median Interquartile Range (IQR) of the Time That it Takes to Complete Visit Number One
Description: Results reflect the time taken to complete visit 1 in minutes. Data was collected using time-stamp data from the Redcap system.
Time Frame: Baseline visit (V1)
Population: 1 participant withdrew prior to starting treatment.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Transcutaneous Electrical Acustimulation (TEA)
Number analyzed (Participants) | 9
minutes | 22 [13 to 56.5]

8. Primary Outcome: Median Interquartile Range (IQR) of the Time That it Takes to Complete Visit Number Two
Description: Results reflect the time taken to complete visit 2 in minutes. Data was collected using time-stamp data from the Redcap system.
Time Frame: 4 weeks (after treatment period)
Population: 1 participant withdrew prior to receiving treatment. 2 participants did not provide data at the second visit, as they did not complete the questionnaires.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Transcutaneous Electrical Acustimulation (TEA)
Number analyzed (Participants) | 7
minutes | 10 [10 to 11]

9. Primary Outcome: Proportion of Participants Who Came for Visit 1 and Completed All the Surveys Involved in the Study
Description: Results reflect the participants who came for visit 1 and completed all the surveys involved in the study.
Time Frame: Approximately 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Transcutaneous Electrical Acustimulation (TEA)
Number analyzed (Participants) | 10
Participants | 0

10. Primary Outcome: Percentage of Study Surveys That Were Completed Per Protocol
Description: Results reflect the percentage of surveys that participants completed during the treatment period (between visit 1 and visit 2) and the follow-up period (between visit 2 and visit 3). Each participant was sent 80 surveys total between visits 1 and 3, with 40 being sent between visit 1 and visit 2, and 40 being sent between visit 2 and visit 3. The time between visit 1 and visit 2 was 4 weeks, and the time between visit 2 and visit 3 was 4 weeks.
Time Frame: 8 weeks
Population: 1 participant withdrew prior to starting treatment, so no survey data was collected.
Measure: Number; unit: percentage of surveys completed
Units Other Than Participants: Surveys
Arm/Group | Transcutaneous Electrical Acustimulation (TEA)
Number analyzed (Participants) | 9
Number analyzed (Surveys) | 720
percentage of surveys completed
  between visit 1 and visit 2 | 71.3
  between visit 2 and visit 3 | 63.2

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Arm/Group | Transcutaneous Electrical Acustimulation (TEA)
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transcutaneous Electrical Acustimulation (TEA) (N=10)
Pneumonia (Infections and infestations) | 1 — One participant withdrew from the trial for an unrelated admission due to pneumonia prior to receiving any TEA session or starting treatment questionnaires.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT06015945/Prot_SAP_000.pdf